CLINICAL TRIAL: NCT00043940
Title: Anticoagulant Therapy With Bivalirudin in the Performance of PCI in Patients With Heparin-Induced Thrombocytopenia
Brief Title: Anticoagulant Therapy With Bivalirudin in the Performance of Percutaneous Coronary Intervention in Patients With Heparin-Induced Thrombocytopenia (AT BAT, First Inning)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMC-98-10
Record Dates: First submitted 2002-08-14; First posted 2002-08-16 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Heparin-Induced Thrombocytopenia; Thrombosis
Keywords: thrombosis; bivalirudin; direct thrombin inhibitor; HIT; HITTS; HIT/HITTS
MeSH Terms: conditions — Thrombosis | interventions — bivalirudin

INTERVENTIONS:
Drug: bivalirudin — Bivalirudin therapy will be given as a 0.75-mg/kg intravenous bolus and 1.75-mg/kg/h intravenous infusion during procedure and up to 4 hours.

SUMMARY:
Primary Objective:

To assess the safety of bivalirudin as an alternative anticoagulant therapy for patients with new or previous heparin-induced thrombocytopenia (HIT) / heparin-induced thrombocytopenia and thrombosis syndrome (HITTS) undergoing percutaneous coronary intervention (PCI). This will be measured by the composite incidence of major bleeding events during administration or within 48 hours after stopping bivalirudin (or at hospital discharge, whichever occurs first). The components of the composite endpoint are: a) intracranial bleeding; b) retroperitoneal bleeding; c) bleeding that results in hemodynamic compromise; d) bleeding that requires transfusion of three or more units of whole blood or packed red cells; and e) a decrease in hemoglobin of greater than or equal to g/dL or in hematocrit of greater than or equal to 9%.

Secondary Objectives:

Each component of the primary composite endpoint.

To evaluate the level of anticoagulation achieved with bivalirudin. The goal is to achieve an activated clotting time (ACT) between 300 and 350 sec during PCI and 4-hour bivalirudin infusion.

To evaluate bivalirudin's effects on platelet counts.

ELIGIBILITY:
INCLUSION:

* Males and females at least 18 years of age,
* Be able to provide written informed consent,
* Need anticoagulation for percutaneous coronary intervention (angioplasty, rotational atherectomy, directional coronary atherectomy, transluminal extraction catheter, or coronary stent),
* New diagnosis or history of clinically suspected or objectively documented HIT/HITTS, defined as:

(A) Positive heparin-induced platelet aggregation (HIPA) or other functional assay, defined as: (B) HIT: Thrombocytopenia associated with heparin therapy, where the platelet count: (i) has decreased to <100x10(9)/L (minimum of 30% drop from the platelet count before heparin treatment), OR (ii) has decreased to <150x10(9)/L (minimum of 40% drop from the platelet count before heparin treatment, OR, (C) HITTS: Thrombocytopenia (as defined above) PLUS arterial or venous thrombosis (deep-vein thrombosis, pulmonary embolism, mesenteric venous or arterial thrombosis, acute myocardial infarction, left ventricular thrombus, ischemic stroke, or occlusion or limb arteries), diagnosed by physical exam/lab evidence and/or appropriate imaging studies (duplex ultrasound, venography, ventilation-perfusion scan, venous or arterial angiography, MRI/MRA, catheterization).

EXCLUSION:

* Overt or known active significant bleeding,
* Definitive evidence of an alternative explanation for the thrombocytopenia (e.g.m DIC, sepsis, other consumptive coagulopathy, ITP, TTP, HUS, or bone-marrow failure),
* Coagulation disorder or bleeding diathesis unrelated to HIT/HITTS,
* Patients with renal impairment, defined as calculated creatinine clearance <30 mL/min, or any other medical conditions (including hepatic, pulmonary, gastrointestinal, endocrine, or psychiatric) that, in the investigator's opinion, would endanger the patient if she/he receives anticoagulant therapy,
* Nonhemorrhagic stroke within the past 6 months or any previous hemorrhagic stroke,
* Intracranial neoplasm, or cerebral/spinal arteriovenous malformation or aneurysm,
* Lumbar puncture, or spinal/epidural catheter placement within the past 7 days,
* Known prior hemorrhage (gastrointestinal, genitourinary, pericardia, pleural, retroperitoneal spaces), major surgery, or serious trauma within the past 6 weeks, unless attending physician believes the need for anticoagulation with PCI outweighs the potential bleeding risk,
* Puncture of a non-compressible vessel within 24 hours before the planned PCI,
* Confirmed uncontrolled hypertension (systolic blood pressure > or = 100 mmHg) at study entry,
* Ongoing anticoagulant therapy at study entry. However, patients may be entered if the therapy can be safely stopped periprocedurally, or, in the case of oral warfarin, if the prothrombin time INR can safely be brought to < or = 1.5 just before study drug infusion,
* Known or suspected pregnancy, or breast-feed. Women of childbearing potential must have a negative pregnancy test (urine or blood) and must be made explicitly aware that bivalirudin may cause excessive menstrual bleeding. Known or suspected pregnancy, or breast-feeding,
* Known hypersensitivity to bivalirudin or leech proteins,
* If the patient has participated in a drug trial within the past 48 hour, call the DCRI hotline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 1999-04; Primary Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Major bleeding events | 48 hours
  composite incidence of major bleeding events during administration or within 48 hours after stopping bivalirudin

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Clinical Research Institute, Duke University Medical Center, Durham, North Carolina, United States